CLINICAL TRIAL: NCT06468709
Title: A Prospective, Randomized Controlled Trial on the Recurrence Free Survival Rate of Type I AIP With High-risk of Recurrence Patients Receiving Glucocorticoid Maintenance Therapy/Glucocorticoid Combined With MMF Maintenance Therapy
Brief Title: A Trial on the Recurrence Free Survival Rate of Type I AIP With High-risk of Recurrence
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, ZOU DUOWU, Director of Gastroenterology Department, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2024-107
Record Dates: First submitted 2024-05-23; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Type 1 AIP
Keywords: Type 1 AIP; Recurrence; Glucocorticoids; MMF
MeSH Terms: conditions — Autoimmune Pancreatitis; Recurrence | interventions — Glucocorticoids; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucocorticoids group (Active Comparator): Induction therapy: Prednisone 30mg/d, lasting for 4 weeks, then decreasing by 5mg/d every 2 weeks until maintained at 5mg/d
  Interventions: Drug: Glucocorticoids
- Glucocorticoids+MMF group (Experimental): GC: Induction therapy: 30mg/d, lasting for 4 weeks, then decreasing by 5mg/d every 2 weeks until maintained at 5mg/d. At the initial stage of simultaneous treatment, 1.0g-1.5g MMF combined with GC treatment
  Interventions: Drug: Glucocorticoids+MMF

INTERVENTIONS:
Drug: Glucocorticoids — The study subjects were randomly divided into a GC monotherapy maintenance group and a GC combined with MMF maintenance group in a 1:1 ratio. The randomization sequence was generated online using a computer randomization scheme. Group A was the GC monotherapy maintenance group
  Other Names: Prednisone
  Arms: Glucocorticoids group
Drug: Glucocorticoids+MMF — The study subjects were randomly divided into a GC monotherapy maintenance group and a GC combined with MMF maintenance group in a 1:1 ratio. The randomization sequence was generated online using a computer randomization scheme. Group B was the GC+MMF maintenance group
  Other Names: Prednisone and MMF
  Arms: Glucocorticoids+MMF group

SUMMARY:
Autoimmune pancreatitis (AIP) is an autoimmune disease with low incidence rate and involving the pancreas. In China, type I AIP is predominant. Glucocorticoids (GC) have a significant therapeutic effect. Even though a consensus has been reached on the effective initial GC treatment dose, type I AIP is prone to recurrence after GC induction and maintenance therapy. Currently, there is no consensus on how to reduce the disease recurrence rate in high-risk type I AIP patients. Multiple studies have shown that immunosuppressants (IM) combined with GC can effectively reduce the disease recurrence rate in IgG4 RD patients, including azathioprine, mycophenolate mofetil (MMF), etc. Among them, the incidence of adverse reactions in MMF is relatively low. As a special type of IgG4-RD, there is currently no prospective study evaluating the efficacy and safety of GC combined with MMF treatment in high-risk recurrent type I AIP patients. The smooth implementation of this project can provide new treatment ideas and evidence-based medicine for reducing the recurrence rate of high-risk type I AIP.

DETAILED DESCRIPTION:
Autoimmune pancreatitis (AIP) is an autoimmune disease with low incidence rate and involving the pancreas. It can be divided into type I AIP and type II AIP. In China, type I AIP is predominant, accompanied by elevated IgG4 levels, diffuse or segmental pancreatic enlargement, and irregular narrowing of the pancreatic duct. Glucocorticoids (GC) have a significant therapeutic effect. Even though a consensus has been reached on the effective initial GC treatment dose, type I AIP is prone to recurrence after GC induction and maintenance therapy. Currently, there is no consensus on how to reduce the disease recurrence rate in high-risk type I AIP patients. The International Pancreatic Society has released an international consensus on AIP, indicating that the risk factors for AIP recurrence are still unclear. The following are possible signs of recurrence: IgG4>4 times the upper limit of normal value before treatment; The serum IgG4 level remained high after GC treatment; Pancreatic diffuse enlargement; IgG4-SC with proximal bile duct involvement; Involvement of extrapancreatic organs.Multiple studies have shown that immunosuppressants (IM) combined with GC can effectively reduce the disease recurrence rate in IgG4 RD patients, including azathioprine, mycophenolate mofetil (MMF), etc. Among them, the incidence of adverse reactions in MMF is relatively low. As a special type of IgG4-RD, there is currently no prospective study evaluating the efficacy and safety of GC combined with MMF treatment in high-risk recurrent type I AIP patients. The smooth implementation of this project can provide new treatment ideas and evidence-based medicine for reducing the recurrence rate of high-risk type I AIP.Main research objective: To evaluate the impact of corticosteroid monotherapy and corticosteroid combined with MMF maintenance therapy on disease remission rate in high-risk type I AIP patients with recurrence within 3 years Secondary research objective: (I) To evaluate the impact on endocrine function; (II) Evaluate the impact on external secretion function; (III) Evaluate the impact on the incidence of malignant tumors; (IV) Adverse reactions; (V) Treatment costs

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form with date;
2. Promise to comply with research procedures and cooperate with the implementation of the entire process research;
3. Age 18 and above, regardless of gender;
4. Confirmed as type I AIP and high-risk for recurrence, including the following characteristics: IgG4>4 times the upper limit of normal value before treatment; The serum IgG4 level remained high after GC treatment; Pancreatic diffuse enlargement; IgG4-SC with proximal bile duct involvement; Involvement of extrapancreatic organs;
5. Indications for treatment, (1) symptomatic individuals may experience pancreatic involvement (such as obstructive jaundice, abdominal pain, lower back pain, etc.) and extrapancreatic organ involvement (such as jaundice caused by bile duct stenosis, etc.); (2) Asymptomatic individuals, who may develop subclinical AIP (persistent pancreatic mass, liver dysfunction with proximal IgG4 associated sclerosing cholangitis) with severe and irreversible damage to important organs;
6. Able to persist and cooperate with research interventions, such as oral medication;
7. If it is a woman in the reproductive period, contraception should be used for at least one month before screening, and a commitment should be made to use contraception throughout the entire study period and continue until the specified time after the end of the study

Exclusion Criteria:

1. Pregnant/lactating women; Inability or refusal to sign informed consent form;
2. History of mental illness;
3. Allergy to research interventions;
4. With malignant tumors;
5. Active hepatitis/tuberculosis and other infectious diseases;
6. With underlying diseases that are difficult to control, such as severe heart failure, respiratory failure, etc;
7. Within 3 months, use of glucocorticoids or immunosuppressants due to other illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the impact of monotherapy with glucocorticoids and glucocorticoid combined with MMF maintenance therapy on disease remission rate in high-risk type I AIP patients for recurrence within 3 years | 3 years
  to evaluate the disease remission rate of monotherapy with glucocorticoids and glucocorticoid combined with MMF maintenance therapy in high-risk type I AIP patients within 3 years

SECONDARY OUTCOMES:
Evaluate the impact on endocrine function | 3 years
  to evaluate the incidence rate of diabetes mellitus, including measuring Hb1Ac, C peptide, insulin secretion.
Evaluate the impact of external secretion pancreatic function | 3 years
  to evaluate the incidence rate of external secretion disfunction of pancreas including the level of vitamin, 25-OH-D3
Assess the impact on the incidence of malignant tumors | 3 years
  to assess the impact on the incidence of gastrointestinal tumors by endoscopies
Adverse reactions | 3 years
  Adverse reactions including the allergic reactions to drugs
Treatment costs | 3 years
  to assess the total treatment costs in 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Duowu Zou, Doctor, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD